CLINICAL TRIAL: NCT00004257
Title: A Phase I Study of Oxaliplatin in Combination With Continuous Infusion 5-Fluorouracil and Radiation in Esophageal Cancer
Brief Title: Oxaliplatin and Fluorouracil Plus Radiation Therapy in Treating Patients With Primary Esophageal or Stomach Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067504; ALB-RPCI-DS-99-08; RPCI-DS-99-08; NCI-T99-0061
Record Dates: First submitted 2000-01-28; First posted 2003-04-18 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2007-12

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Fluorouracil; Oxaliplatin; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: oxaliplatin
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug and combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining oxaliplatin and fluorouracil plus radiation therapy in treating patients who have primary esophageal or stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of oxaliplatin when given in combination with continuous-infusion fluorouracil and radiotherapy in patients with primary cancer of the thoracic esophagus or gastroesophageal junction.
* Determine the pharmacokinetics of this regimen in this patient population.
* Assess somatic p53 mutations in cancer of the esophagus and determine their relation to therapeutic response induced by this regimen.
* Assess, in a preliminary manner, the efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study of oxaliplatin and fluorouracil.

Patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29 and fluorouracil IV continuously on days 8-42. Patients also undergo radiotherapy once daily, 5 days a week, for 6 weeks beginning on day 8.

Patients without evidence of distant disease or unresectable local regional invasion undergo esophageal resection between days 63-70 (within 3-4 weeks after completion of chemoradiotherapy). Patients then receive oxaliplatin as above on days 105, 119, and 133 and fluorouracil as above on days 105-147.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin and fluorouracil until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 4 weeks.

PROJECTED ACCRUAL: A total of 56 patients will be accrued for this study within approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (below 20 cm from incisors) or gastroesophageal (GE) junction

  * Stage I-III
  * Bronchoscopy with biopsy and cytology required if primary esophageal cancer is less than 26 cm from incisors
* No disease outside esophagus and peri-esophageal soft tissue
* GE junction tumors must be confined to no greater than 2 cm into the gastric cardia
* Supraclavicular lymph nodes at station 1 must be less than 1.5 cm or nonpalpable by physical examination

  * Nodes 1.5 cm or greater or palpable by physical examination must be confirmed to be nonmalignant by biopsy
* Subdiaphragmatic lymph nodes at stations 15-20 must be no greater than 1.5 cm
* No recurrent disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm3
* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No grade 2 peripheral neuropathy
* No history of allergy to platinum compounds
* No history of allergy to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No other malignancy within the past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No colony-stimulating factor therapy during first study course

Chemotherapy:

* No prior chemotherapy for esophageal cancer
* At least 4 weeks since other prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for esophageal cancer
* At least 4 weeks since other prior radiotherapy

Surgery:

* No prior resection or attempted resection of esophageal cancer

Other:

* No other concurrent investigational drugs
* No other concurrent commercial agents or therapies for esophageal cancer
* No concurrent highly active antiretroviral agents (HAART) for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P. Leichman, MD, Study Chair — Albany Medical College
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Background] Smith PF, Booker B, Pendyala L, et al.: Pharmacokinetic modeling of oxaliplatin with and without 5-FU and radiation. [Abstract] Proc Am Assoc Cancer Res 42: A-2913, 542, 2001.
- [Result] Khushalani N, Nava H, Leichman CG, et al.: A phase I study of oxaliplatin in combination with continous infusion 5-fluorouracil and radiation in esophagus cancer. [Abstract] Proc Am Assoc Cancer Res 42: A-3751, 697, 2001.
- [Result] Pendyala L, Leichman CG, Clark K, et al.: Oxaliplatin, 5-fluorouracil, and radiation in cancer of the esophagus: a pharmacokinetic (PK)/molecular correlates study. [Abstract] Proc Am Assoc Cancer Res 42: A-3347, 623, 2001.